CLINICAL TRIAL: NCT03087760
Title: Phase II Trial of Consolidation Pembrolizumab After Concurrent Chemotherapy and Proton Reirradiation for Thoracic Recurrences of Non-Small Cell Lung Cancer
Brief Title: Trial of Consolidation Pembrolizumab After Concurrent Chemotherapy and Proton Reirradiation for Thoracic Recurrences of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 16516
Record Dates: First submitted 2017-03-17; First posted 2017-03-22 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single Arm, Open Label
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Concurrent Pembrolizumab after proton reirradiation

SUMMARY:
The main purpose of this study is to assess the safety, tolerability and anti-tumor activity of the experimental study drug pembrolizumab (also known as Keytruda or MK-3475) in people with non-small cell lung cancer (NSCLC) that has come back after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of NSCLC who have received previous intrathoracic radiation therapy with definitive intent and have a tumor recurrence in or near the prior irradiation fields. Re-biopsy of the recurrence is not required and is left to the discretion of the treating physician, although every effort should be made to confirm recurrence pathologically.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Age 18 or greater
* Patients with prior invasive malignancies are allowed, provided they have been treated with definitive intent and have no evidence of active disease requiring treatment in the past 2 years.
* Patients must be capable of giving informed consent and be willing and able to comply with schedule.
* Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN.
* Platelets >100,000 cells/mm3 and ANC > 1,250 cells/mm3
* Creatinine ≤ 1.5 X ULN OR measured or calculated creatinine clearance ≥50 mL/min for subject with creatinine levels > 1.5 X institutional ULN. (GFR can also be used in place of creatinine or CrCl).
* Clinical target volume (CTV) size must be <250 cc, no more than 74 Gy of prior radiation in 2 Gy fractions previously administered.

Exclusion Criteria:

* Allergy to Pembrolizumab or related compounds
* History of symptomatic CTCAEv4 grade ≥3 pneumonitis following the initial course of definitive radiation therapy
* History of symptomatic idiopathic pulmonary fibrosis or interstitial lung disease
* Use of continuous oxygen
* Diagnosis of immunodeficiency or exposure to systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. (Nasal or oral inhalers are permissible).
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome are not excluded from the study.
* History of allogenic tissue or solid organ transplant
* Progression while on prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Patients with known extrathoracic metastases, including brain metastases, or known malignant pleural or pericardial effusion
* Prior radiation treatment less than 6 months from the planned start of reirradiation of any part of the intended treatment volume
* Pregnant or breast-feeding patients. Men and women of reproductive potential may not participate in this study unless they have agreed to use an effective contraceptive method while in this study.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg positive or HBV DNA detectable) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feigenberg, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Yegya-Raman N, Berman AT, Ciunci CA, Friedes C, Berlin E, Iocolano M, Wang X, Lai C, Levin WP, Cengel KA, O'Reilly SE, Cohen RB, Aggarwal C, Marmarelis ME, Singh AP, Sun L, Bradley JD, Plastaras JP, Simone CB 2nd, Langer CJ, Feigenberg SJ. Phase 2 Trial of Consolidation Pembrolizumab After Proton Reirradiation for Thoracic Recurrences of Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2024 May 1;119(1):56-65. doi: 10.1016/j.ijrobp.2023.08.047. Epub 2023 Aug 29. PMID 37652303
- See also: Phase II trial of consolidation pembrolizumab after proton reirradiation for thoracic recurrences of non-small cell lung cancer: Pembro after PBT ReRT for NSCLC — https://doi.org/10.1016/j.ijrobp.2023.08.047

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between November 2017 and April 2021, 32 patients were consented and reviewed for eligibility, of which 10 were excluded. Most common reasons for exclusion were internal clinical target volume (iCTV) ≥250 cc on the simulation scan (n = 3), histology other than non-small cell lung cancer (NSCLC) (n = 3), and extrathoracic metastases (n = 2). Twenty-two patients initiated proton beam therapy (PBT) reirradiation (reRT) on-trial and were included in the intention-to-treat analysis.
Groups:
- Single Arm: Single Arm, Open Label
  Pembrolizumab 100 mg/4mL (dosage form: solution for injection). Pembrolizumab will be administered as a 30 minute intravenous infusion. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).
  Concurrent Pembrolizumab after proton reirradiation.
Period: Overall Study
Arm/Group | Single Arm
Started | 22
Completed | 3
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 68 [54 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 1
  Unknown or Not Reported | 1
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — The investigator or qualified designee will assess ECOG status at screening, prior to the administration of each dose of trial treatment and discontinuation of trial treatment as specified in the Trial Flow Chart.
  Grade 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    Eastern Cooperative Oncology Group (ECOG) performance status: 0 | 7
    Eastern Cooperative Oncology Group (ECOG) performance status: 1 | 15
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 12
  Squamous cell carcinoma | 8
  Adenosquamous | 1
  Non-small cell lung cancer (NSCLC), not otherwise specified | 1
Programmed death-ligand (PD-L1 ) [Count of Participants; unit: Participants]
  <1% | 9
  1-50% | 9
  >50% | 3
  Not Applicable (N/A) | 1
Epidermal growth factor receptor (EGFR) mutation [Count of Participants; unit: Participants] | 1
Anaplastic lymphoma kinase (ALK) translocation [Count of Participants; unit: Participants] | 1
Recurrence location [Count of Participants; unit: Participants]
  Primary tumor | 4
  Nodal | 8
  Primary tumor + nodal | 10
Prior overlapping radiation therapy - Definitive chemoradiation [Count of Participants; unit: Participants] — Population: 15 out 22 participants had prior overlapping radiation therapy - definitive chemoradiation.
  Participants
    number analyzed (Participants) | 15
    Intensity modulated radiation therapy (IMRT) | 11
    Passive scatter proton beam therapy (PBT) | 2
    Pencil beam scanning proton beam therapy (PBT) | 2
Prior overlapping radiation therapy - Stereotactic body radiation therapy (SBRT) [Count of Participants; unit: Participants] | 3
Prior overlapping radiation therapy - Pre-operative chemoradiation (IMRT) [Count of Participants; unit: Participants] | 1
Prior overlapping radiation therapy - Post-operative chemoradiation (3D-CRT) [Count of Participants; unit: Participants] — Three Dimensional Conformal Radiation Therapy (3D-CRT)
  Participants | 1
Prior overlapping radiation therapy - Definitive chemoradiation (passive scatter PBT) and SBRT [Count of Participants; unit: Participants] | 1
Prior overlapping radiation therapy - Pre-operative (IMRT) and post-operative (IMRT) chemoradiation [Count of Participants; unit: Participants] | 1
Prior surgery for lung cancer [Count of Participants; unit: Participants] — Population: 8 out of the 22 analyzed participants had prior surgery for lung cancer.
  Participants
    number analyzed (Participants) | 8
    Lobectomy | 6
    Wedge resection | 2
Prior consolidation durvalumab [Count of Participants; unit: Participants] | 8
Prior consolidation durvalumab - Median duration [Median (Full Range); unit: months] | 12 [7 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Progression Free Survival
Description: Progression Free Survival is defined as the time from initiation of definitive therapy to the first documented disease progression per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 based on radiologists' review or death due to any cause, whichever occurs first, or last patient follow-up that documented lack of disease progression. Patients who have not had disease progression or who have died, will be censored on the most recent clinical evaluation date that documented that they were progression-free.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 22
Participants | 6

2. Secondary Outcome: Number of Participants Who Experienced a Grade 3+ Adverse Event
Description: Toxicity was graded using the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0. Adverse events were reviewed by the treating physicians and principal investigator to assess potential attribution to reirradiation/chemotherapy or pembrolizumab.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 22
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events will be monitored during Pembrolizumab treatment and for one year following treatment for patients who completed all 17 cycles of Pembrolizumab, up to 2 years.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 14/22
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=22)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 3
Tracheal rupture (Injury, poisoning and procedural complications) | 1
Aorto-esophageal fistula (Gastrointestinal disorders) | 1
Recurrent Laryngeal Nerve Damage (Respiratory, thoracic and mediastinal disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Oral mucositis and lichenoid dermatitis (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=22)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Weakness (Musculoskeletal and connective tissue disorders) | 1
Gastroesopheal reflux (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Leg edema (General disorders) | 1
Myalgia or arthralgia (Musculoskeletal and connective tissue disorders) | 3
Elevated BUN (Blood and lymphatic system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hyperthyroidism (Endocrine disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Elevated creatinine (Investigations) | 1
Neuropathy (Nervous system disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 5
Hypothyroidism (Endocrine disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/60/NCT03087760/Prot_SAP_000.pdf